CLINICAL TRIAL: NCT05187013
Title: mHealth to Address Uncontrolled Hypertension Among Hypertensive Homeless Adults
Brief Title: Uncontrolled Hypertension Among the Homeless
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: New York University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Ramin Asgary, Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCR203140; 1R21MD016201-01 (NIH)
Record Dates: First submitted 2021-12-07; First posted 2022-01-11 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Hypertension
Keywords: Hypertension; Homeless Persons; mHealth; Short message service; texting; blood pressure; medication adherence
MeSH Terms: conditions — Hypertension; Medication Adherence | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertension-Specific Education (Experimental): 6 months of mHealth HTN management support via SMS texts including reminders for medication adherence, appointment attendance, and HTN-specific health education and support. Texts will be delivered to support medication adherence and lifestyle changes, and participants will receive appointment reminders before each appointments with a follow-up text and robocall if the appointment is missed.
  Interventions: Behavioral: mHealth for Hypertension in Homeless Persons
- General Health Education (Other): 6 months of mHealth including basic healthcare and general health promotion via SMS texts. Blood pressure measurements and adherence assessments will be collected at every shelter visit.
  Interventions: Behavioral: mHealth for Hypertension in Homeless Persons

INTERVENTIONS:
Behavioral: mHealth for Hypertension in Homeless Persons — SMS text messages sent to participants' mobile phones

SUMMARY:
This study is designed to assess the effect of implementing a mobile health (mHealth) strategy using text messaging for hypertension (HTN) management among hypertensive homeless persons with uncontrolled blood pressure age 21 or older in shelter-clinics in New York City (NYC). The study uses a randomized clinical trial design (homeless, n=120) and semi-structured interviews (homeless, n=30; providers, n=20).

The control group will receive text messages for usual standard care/healthy lifestyle during a 6-month follow-up period. The intervention group will receive text messages geared towards both standard care/healthy lifestyle and blood pressure control. At the end of study period, the investigators will assess changes in blood pressure (BP) measurements, adherence to clinic visits, and adherence to medication, and the investigators will compare them between the two groups. Qualitative interviews with both patients and providers who provide services to the homeless in shelter settings will develop a better understand barriers and opportunities regarding BP control. The investigators hypothesize that those individuals randomized to the intervention will experience a reduction in blood pressure (8mmHg systolic BP or diastolic BP) and will exhibit better adherence to blood pressure medications and appointments compared to the control group.

DETAILED DESCRIPTION:
Project Renewal operates several urban shelters in five boroughs of NYC. Enrollment, data collection, and retention will be supported at these sites.

Patient participants will be recruited in clinics via medical record reviews and will be randomly assigned to treatment groups using a computer-assisted permuted randomization schedule with a block size of four, stratified by clinic site, severe mental illness, and active substance use disorder. Provider participants are physicians, nurse practitioners, social workers, and counselors working at Project Renewal.

The intervention will include 6 months of mHealth HTN management support via short message service (SMS) texts including reminders for medication adherence, appointment attendance, and HTN-specific health education and support. Texts will be delivered to support medication adherence and lifestyle changes, and participants will receive appointment reminders before each appointments. The control group will receive 6 months of mHealth including basic healthcare and general health promotion via SMS texts on the same schedule as the intervention group. Both groups will undergo BP measurements and adherence assessments at appointments in the shelter-clinics. All texts will be interactive and reciprocal; during the study, feedback to SMS texts, including automated and reciprocal feedback for patient-specific input, will be directly provided to patients to enhance education and behavioral changes.

Primary outcome measures will be recorded at 0, 2, 4, and 6 months, and secondary outcome measures will be collected throughout the study. Qualitative interviews with persons experiencing homelessness with HTN (n=30, 15 each arm) and providers (n=20) will be conducted at the end of the recruitment period. Trained research assistants (RA) will collect data and perform the semi-structured interviews.

During clinic visits, BP will be measured by trained clinic nurses in a seated upright position on the right arm with a properly sized cuff. Two readings will be taken at 2-minute intervals following 5 minutes of rest and will be averaged and recorded. Proportion of days covered (PDC) and pill counts will be conducted at each visit. Additional information, including appointment attendance, will be collected from the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing homelessness
* Current diagnosis of hypertension
* SBP above 140mmHg or DBP above 90mmHg at most recent clinic visit
* English or Spanish speaking
* Currently presenting to Project Renewal shelter-clinics for medical care
* Connected to multidisciplinary social and health services at Project Renewal

Exclusion Criteria:

* Pregnant or within 3 months post-partum
* Heart attack or stroke within previous 6 months
* History of aortic aneurysm
* Diagnosis of end-stage renal disease or currently on dialysis
* Inability to read or respond to SMS texts
* Any condition preventing participants from providing informed consent
* SBP >175mmHg or DBP >105mmHg unless medical provider determines patient has no symptoms suggesting a hypertensive emergency or urgency

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Asgary, MD, MPH, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Asgary R, Bauder L, Naderi R, Ogedegbe G. SMS text intervention for uncontrolled hypertension among hypertensive homeless adults in shelter clinics of New York City: protocol for a pragmatic randomised trial study. BMJ Open. 2023 Oct 30;13(10):e073041. doi: 10.1136/bmjopen-2023-073041. PMID 37903607

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant study events occurred after participant enrollment and before study assignment.
Groups:
- Providers: Healthcare providers who participated in the semi-structured interview only.
Period: Overall Study
Arm/Group | Hypertension-Specific Education | General Health Education | Providers
Started | 57 | 56 | 10
Number of Individuals Who Participated in Semi-Structured Interviews | 13 | 7 | 10
Completed | 33 | 32 | 10
Not Completed | 24 | 24 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 20 | 17 | 0
Not completed — Ongoing Participants | 3 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Providers only participated in semi-structured interviews. No baseline or demographic data were collected for this group.
Groups:
- Providers: Healthcare providers and shelter staff who participated only in semi-structured interviews. No demographic data was collected for this group.
- Total: Total of all reporting groups
Arm/Group | Hypertension-Specific Education | General Health Education | Providers | Total
Number analyzed (Participants) | 57 | 56 | 0 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.53 (10.2) | 58.05 (9.66) |  | 57.78 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 |  | 11
  Male | 51 | 51 |  | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 |  | 1
  Asian | 1 | 1 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 |  | 2
  Black or African American | 38 | 33 |  | 71
  White | 7 | 5 |  | 12
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 11 | 14 |  | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 16 |  | 30
  Not Hispanic or Latino | 42 | 35 |  | 77
  Unknown or Not Reported | 1 | 5 |  | 6
Blood Pressure Baseline, Systolic, and Diastolic [Mean (Standard Deviation); unit: mmHG] — Baseline values for participants' blood pressure values, both systolic and diastolic
  mmHG
    Systolic Blood Pressure | 155.772 (12.071) | 156.018 (11.771) |  | 155.894 (11.871)
    Diastolic Blood Pressure | 91.263 (10.316) | 93.482 (11.323) |  | 92.363 (10.836)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: Systolic and diastolic blood pressure readings (SBP and DBP)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Hypertension-Specific Education | General Health Education
Number analyzed (Participants) | 33 | 32
mmHG
  Systolic Blood Pressure | 135.36 (18.31) | 136.19 (15.68)
  Diastolic Blood Pressure | 89.67 (10.71) | 92.38 (82.22)
Statistical Analysis 1: Comparison: Hypertension-Specific Education vs General Health Education; Null Hypothesis: No improvement between baseline and final SBP, i.e., Final SBP - Baseline SBP >= 0 Alternative Hypothesis: Final SBP - Baseline SBP <0 Power calculation: Based on the data, the mean and SD of the change in SBP are -7.16 and 21.40, respectively. Using a one-sided paired t-test with a significance level of 0.05, we should have a power of 83.16%; Test type: Superiority; p = 0.006, t-test, 1 sided; Mean Difference (Net) = -7.16, 95% CI 2-sided [-12.59 to -1.73], Standard Error of Mean 2.72
Statistical Analysis 2: Comparison: Hypertension-Specific Education vs General Health Education; Null Hypothesis: No improvement between baseline and final DBP, i.e., Final DBP - Baseline DBP >= 0 Alternative Hypothesis: Final DBP - Baseline DBP <0 Power calculation: Based on the data, the mean and SD of the change in SBP are -2.15 and 10.49, respectively. Using a one-sided paired t-test with a significance level of 0.05, we should have a power of 51.48%; Test type: Superiority; p = 0.056, t-test, 1 sided; Mean Difference (Net) = -2.15, 95% CI 2-sided [-4.79 to 0.49], Standard Error of Mean 1.32
Statistical Analysis 3: Comparison: Hypertension-Specific Education vs General Health Education; Null hypothesis: No difference between the change in SBP between the two arms Power calculation: With our sample size, we expect to have 80% power as long as the effect size is at least 0.72 at a 5% level; Test type: Equivalence — The margin was considered to be 0; p = 0.87, ANCOVA; Adjusted for baseline SBP and follow-up time; Mean Difference (Net) = -0.67, 95% CI 2-sided [-8.76 to 7.42], Standard Error of Mean 4.13 — The parameter was defined as the change in SBP for the general health education arm - the change in SBP for the HTN specific education arm adjusted for follow-up time and baseline SBP
Statistical Analysis 4: Comparison: Hypertension-Specific Education vs General Health Education; Null hypothesis: No difference between the change in DBP between the two arms Power calculation: With our sample size, we expect to have 80% power as long as the effect size is at least 0.72 at a 5% level; Test type: Equivalence — The margin was taken to be 0; p = 0.63, ANCOVA; Adjusted for baseline DBP and follow-up time; Mean Difference (Net) = 0.98, 95% CI 2-sided [-3.02 to 4.98], Standard Error of Mean 2.04 — The parameter was defined as the change in DBP for the general health education arm - the change in DBP for the HTN specific education arm adjusted for follow-up time and baseline SBP

2. Primary Outcome: Medication Adherence
Description: Medication adherence was measured using the Voils 3-Item DOSE-Nonadherence measure, a 5-item Likert scale. This was measured by dichotomizing the response options such that any score of 2-5 on any of the three Extent of Non-adherence items is considered non-adherent (e.g., code as 1), and a response of 1 (none of the time) on all items is considered adherent (e.g., code as 0). The extent of adherence was then reported as a median percentage of the total participants with an IQR range as reflected below.
Time Frame: Overall over 6 months
Measure: Median (Inter-Quartile Range); unit: Percentage of Adherent Participants
Arm/Group | Hypertension-Specific Education | General Health Education
Number analyzed (Participants) | 33 | 32
Percentage of Adherent Participants | 83.3 [25 to 100] | 50 [0 to 100]
Statistical Analysis 1: Comparison: Hypertension-Specific Education vs General Health Education; Null hypothesis: There is no difference in medicine adherence between the two groups; Test type: Equivalence — The margin is taken to be 0; p = 0.14, Regression, Logistic; A mixed effect model with study arm as a fixed effect and subject-specific random effect; Odds Ratio, log = 0.89, 95% CI 2-sided [-0.26 to 2.29], Standard Error of Mean 0.61 — For OR: the general education arm was taken as the baseline (denominator)

3. Primary Outcome: Appointment Attendance
Description: Percentage of appointments attended
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Hypertension-Specific Education | General Health Education
Number analyzed (Participants) | 33 | 32
Percentage | 46.08 (35.81) | 57.41 (33.51)
Statistical Analysis 1: Comparison: Hypertension-Specific Education vs General Health Education; Null hypothesis: No difference in appointment adherence between the study arms; Test type: Equivalence — The margin was taken to be 0; p = 0.32, Regression, Logistic; Binomial regression for appointment attended/appointment scheduled; Odds Ratio, log = -0.19, 95% CI 2-sided [-0.58 to 0.19], Standard Error of Mean 0.20 — The baseline (denominator) was taken to be the general education arm

4. Secondary Outcome: Number of Participants Who Completed Interviews
Description: The number of interviews that were completed concerning participants' experiences.
  All data obtained are qualitative.
Time Frame: 6 months
Population: The number of participants interviewed from each group is below.
Measure: Number; unit: Participants who Completed Interviews
Groups:
- Providers: Healthcare providers and shelter staff who participated only in semi-structured interviews.
Arm/Group | Hypertension-Specific Education | General Health Education | Providers
Number analyzed (Participants) | 33 | 32 | 10
Participants who Completed Interviews | 13 | 6 | 10

ADVERSE EVENTS:
Time Frame: From enrollment to the completion of the Intervention period, up to 6 Months.
Description: One participant died during the study period; this death was unrelated to the intervention.
Groups:
- Providers: Healthcare providers and shelter staff who participated only in semi-structured interviews. No adverse event data were collected for this group.
Arm/Group | Hypertension-Specific Education | General Health Education | Providers
All-Cause Mortality (participants affected / at risk) | 0/57 | 1/56 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56 | 0/10
Other Adverse Events (participants affected / at risk) | 0/57 | 0/56 | 0/10

LIMITATIONS AND CAVEATS:
We faced some challenges with enrollment due to post-pandemic constraints and the unexpected influx of newcomers into the shelter system in New York City, which were later resolved, and we added another enrollment site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT05187013/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT05187013/SAP_001.pdf
  • Informed Consent Form: Patient Informed Consent Form (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT05187013/ICF_002.pdf
  • Informed Consent Form: Provider Informed Consent Form (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT05187013/ICF_003.pdf